CLINICAL TRIAL: NCT03447977
Title: The Effect of Manual Treatment on Respiratory Parameters, Pain, Posture and Quality of Life in Chronic Neck Pain Individuals
Brief Title: The Effect of Manual Treatment on Respiratory Parameters, Pain, Posture and Quality of Life in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SEVAL TAMER, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-17109
Record Dates: First submitted 2017-12-22; First posted 2018-02-27 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2018-06

CONDITIONS: Neck Pain
Keywords: neck pain; manual therapy; respiratory function
MeSH Terms: conditions — Neck Pain; Respiratory Aspiration | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cervical group (Experimental): cervical spinal mobilizations, exercises, 2 session for 6 weeks
  Interventions: Other: cervical; Other: exercises
- thoracic group (Experimental): cervical and thoracic spinal mobilizations, exercises, 2 session for 6 weeks
  Interventions: Other: cervical; Other: thoracic; Other: exercises
- exercise group (Experimental): exercises, 2 session for 6 weeks
  Interventions: Other: exercises

INTERVENTIONS:
Other: cervical — cervical spine manual therapy
  Other Names: cervical spine mobilization
  Arms: cervical group; thoracic group
Other: thoracic — thoracic spine manual therapy
  Other Names: thoracic spine mobilizations
  Arms: thoracic group
Other: exercises — exercises for pain

SUMMARY:
Neck pain which is common musculoskeletal system problem in all populations, negatively affects functional status and quality of life. Muscle spasms, postural problems in cervical and thoracic regions and impairment on respiratory parameters (respiratory functions and respiratory muscle strength) is seen with neck pain. Manual therapy and exercise are widely preferred in the treatment of neck pain for improve pain, posture, muscle strength, range of motion, functional status and quality of life.

There are some studies showing that manual therapy improves respiratory parameters in pulmonary diseases but studies are lacking for neck pain. Our aim is to indicate that effects of manual therapy, manual therapy for different regions (cervical and/or thoracal region) and exercises for pain, posture, quality of life and also respiratory parameters in patients with chronic neck pain.

DETAILED DESCRIPTION:
Manual therapy and exercises are evidence-based methods for improving pain, muscle strength, range of motion, function and quality of life in individuals with neck pain. These physiotherapy approaches have been shown to improve respiratory functions in patients with neck pain and also in pulmonary diseases such as cystic fibrosis and chronic obstructive pulmonary diseases.

Studies show that to improve respiratory parameters in patients for chronic neck pain, mobilization of thoracic region and exercises for endurance of deep neck muscles are beneficial. Despite the proposal given in this study, there are few studies evaluating the relationship between respiratory functions and the strength of respiratory muscles in patients with neck pain in detail, and also the effectiveness of different physiotherapy-rehabilitation methods on respiratory functions on neck pain. In a single study on this subject, thoracic region manual therapy, stretching exercise program and both of these applications were applied for the subjects. At the end of the treatment, respiratory functions developed in all three groups; but both applications group have been shown to more effective than thoracic manual therapy group for increasing respiratory functions.Exercises and manual therapy for cervical and/or thoracic region frequently used for chronic neck pain but there are no studies that compare manual therapy for different region on respiratory parameters. Therefore, our aim is to determine the effects of exercises with manual therapy methods for cervical and/or thoracic region in chronic neck pain patients on pain, posture, quality of life, as well as on respiratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have pain for at least 3 month with mechanical neck pain
* Individuals voluntarily participating to the study

Exclusion Criteria:

* Individuals who have undergone cervical, spinal, thoracic, or abdominal region surgeries or pathology; whiplash injury; neurological deficit; osteoporosis; rheumatological disease; pulmonary disease; pharmacological treatment; or malignancy; or have a body mass index (BMI) >40 or were smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
respiratory function(forced vital capacity,peak expiratory flow,maximum voluntary ventilation,forced expiratory flow at 1sn) | change from baseline respiratory parameters at six weeks
  respiratory function will be measured with spirometer (%)high degrees represent better outcome, low degrees represent worse outcome)
respiratory muscle strength | change from baseline respiratory muscle strength at six weeks
  inspiratory muscle strength and expiratuary muscle strength will be measured with digital mouth pressure measuring device (%).

SECONDARY OUTCOMES:
pain position | change from baseline pain at six weeks
  pain level at rest, activity and night with visual analog scale (min 0cm-max10cm, better outcome 0 worst outcome 10)
posture | change from baseline posture at six weeks
  forward head posture(high degrees represent worse outcome, low degrees represent better outcome), thoracic posture (high degrees represent worse outcome, low degrees represent better outcome)
range of motion | change from baseline range of motion at six weeks
  neck range of motion(high degrees represent better outcome, low degrees represent worse outcome
neck functional status | change from baseline functional status at six weeks
  neck disability index (total score min 0- max 50 point, high degrees represent worse outcome, low degrees represent better outcome and 0-4 point= no disability, 5-14 minimal disability, 15-24 moderate disability, 25-34 severe disability, 35-50 total functional disability)
quality of life status | change from baseline quality of life at six weeks
  Short form of quality of life scale(SF-36)(total score 100 point min 0-max 100 point, high degrees represent better outcome, low degrees represent worse outcome
anxiety level | change from baseline anxiety level at six weeks
  back anxiety scale(min 0-max 63 point, high degrees represent worse outcome, low degrees represent better outcome, total score 0-17 point shows minimal anxiety, 18-24 shows moderate anxiety, 30-63 shows severe anxiety status)
depression level | change from baseline depression level at six weeks
  back depression scale(min 0-max 63 point,high degrees represent worse outcome, low degrees represent better outcome, total score 0-9 shows minimal depression, 10-16 shows mild depression, 17-29 shows moderate depression, 30-63 shows severe depression status
physical activity level | change from baseline physical activity level at six weeks
  international physical activity score ( the metabolic equivalent (MET) value will be calculated and recorded by asking the time and frequency spent on sitting, walking, moderately severe activities and violent activities. The total physical activity value will be determined using the formula calculated by the patient's body weight, total score < 600 MET-dk/week shows physically inactivity, 600-3000 MET-dk/week shows minimal active and > 3000 MET-dk/week shows active
kinesiophobia | change from baseline kinesiophobia at six weeks
  tampa kinesiophobia scale (total score min 17-max 68 point, high degrees represent worse outcome, low degrees represent better outcome)
neck muscle endurance | change from muscle endurance baseline at six weeks
  The measurements were performed from a crook lying position with a pressure biofeedback device (Stabilizer, Chattanooga, USA), which was placed behind participants' neck. The device was initially inflated to a baseline pressure of 20 mmHg. The participants had to successively perform 3 10-s holds of a head nodding action at each of the 5 pressure levels (22 mmHg, 24 mmHg, 26 mmHg, 28 mmHg and 30 mmHg). Participants' deep neck flexors were considered fatigued when pressure decrease at the pressure sensor, apparent activation of the superficial neck flexors or a jerky action during holding of the pressure level were observed.
neck and upper limb strengths test | change from baseline strength at six weeks
  neck and upper limb strengths test measured with dynamometer (high degrees represent better outcome, low degrees represent worse outcome)
pressure pain | change from baseline strength at six weeks
  pressure pain tolerance with algometer (kg/cm2high degrees represent better outcome, low degrees represent worse outcome
Thoracal expansion | change from baseline expansion strength at six weeks
  the difference between the values obtained during deep inspiration and expiration will be determined by tape (cm),high degrees represent better outcome, low degrees represent worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Seval Tamer, Mcs, Principal Investigator — Hacettepe University Physiotherapy and Rehabilitation
Locations (1):
- Seval Tamer, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 8 months after publication
Access Criteria: requestors will be required to sign a data access agreement

REFERENCES:
- [Background] Hwangbo PN, Hwangbo G, Park J, Lee S. The Effect of Thoracic Joint Mobilization and Self-stretching Exercise on Pulmonary Functions of Patients with Chronic Neck Pain. J Phys Ther Sci. 2014 Nov;26(11):1783-6. doi: 10.1589/jpts.26.1783. Epub 2014 Nov 13. PMID 25435700
- [Background] Wirth B, Amstalden M, Perk M, Boutellier U, Humphreys BK. Respiratory dysfunction in patients with chronic neck pain - influence of thoracic spine and chest mobility. Man Ther. 2014 Oct;19(5):440-4. doi: 10.1016/j.math.2014.04.011. Epub 2014 Apr 30. PMID 24835338
- [Background] Kapreli E, Vourazanis E, Strimpakos N. Neck pain causes respiratory dysfunction. Med Hypotheses. 2008;70(5):1009-13. doi: 10.1016/j.mehy.2007.07.050. Epub 2007 Oct 23. PMID 17959320